CLINICAL TRIAL: NCT06498466
Title: EFFECT OF MYOFASCIAL RELEASE THERAPY IN PATIENTS WITH CERVICAL MYOFASCIAL PAIN SYNDROME
Status: Completed | Type: Observational
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Elzem Bolkan Günaydın, Principal investigator, Ufuk University
Other Study IDs: 12024861-88
Record Dates: First submitted 2024-07-01; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Myofacial Pain Syndromes
MeSH Terms: conditions — Facial Neuralgia | interventions — Myofascial Release Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: myofascial release — Myofascial release therapy (MRT) is a manual therapy technique that involves gradual stretching by a therapist or the individual, acting on the muscles and surrounding fascia. Its effects include increasing joint range of motion and mobility of soft tissues, eliminating imbalances in muscle tone, reducing muscle pain, reducing stress on joints, and increasing neuromuscular efficiency.

SUMMARY:
Objectives: To investigate the effects of myofascial release therapy (MRT) on pain, number of trigger points (TP), pressure pain threshold (PPT), cervical range of motion (ROM), neck disability, and quality of life in the neck pain due to cervical myofascial pain syndrome (MPS).

In this prospective study, patients in Group I (n=30) underwent a standard physical therapy program. Patients in Group II (n=30) additionally underwent MRT 3 days a week. Before and on the 15th day after treatment, patients' pain was measured by visual analog scale (VAS), TP numbers by palpation, PPTs by pressure algometer, cervical ROM by goniometer, disability by Neck Disability Index (NDI) and quality of life by Nottingham Health Profile (NHP) was evaluated.

ELIGIBILITY:
Inclusion Criteria:

* volunteer patients between the ages of 18-65 who complained of neck pain lasting more than 1 month and met the Travell and Simons criteria for the diagnosis of Myofascial pain syndrome

Exclusion Criteria:

* presence of known infectious, inflammatory, tumoral, and advanced degenerative diseases that may cause neck pain, presence of pain reflected from internal organs, history of spine or shoulder fracture or surgery, presence of nerve root involvement findings due to cervical discopathy, having a history of neck manipulation or invasive procedures in the last 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 60 volunteer patients between the ages of 18-65 who complained of neck pain lasting more than 1 month and met the Travell and Simons criteria for the diagnosis of Myofascial pain syndrome.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | 2 weeks
  The patients were asked to mark the severity of their neck pain at rest and with movement on a 10-centimeter (cm) line on the 1st and 15th days (0: minimum 10: maximum). The higher the measured value, the greater the pain intensity.
Trigger Point Numbers | 2 weeks
  In order to detect the trigger points, the neck and back regions of the patients were evaluated by palpation by the physician.
Pressure Pain Threshold | 2 weeks.
  Pressure pain threshold (PPT) was measured with a pressure algometer (Commander[JTECH medical]). The disc head of the pressure algometer was placed on the trigger point at a 90° angle. Before the application, the patient was asked to describe the pain when he/she first felt it.
Cervical Joint Range of Motion (ROM) | 2 weeks
  Cervical ROM measurements were evaluated actively and passively with a goniometer.
Neck Disability Index | 2 weeks
  Disability was evaluated with the Neck Disability Index. This questionnaire, which evaluates subjective symptoms and daily living activities, consists of a total of 10 sections (pain intensity, personal care, lifting, reading, headache, concentration, work life, driving, sleep, and leisure activities).
Nottingham Health Profile | 2 weeks
  Quality of life was assessed with the Nottingham Health Profile. The scale consists of two parts. The first part consists of a total of 38 items, where each item is answered yes or no. This section has a total of 6 sub-dimensions: pain, emotional reactions, sleep, social isolation, physical activity, and energy. The second part consists of 7 items that question whether there are problems in business life, housework, social life, interpersonal relationships, sexual life, hobbies, and holidays, which are the areas of daily life that are most likely to be affected due to the person's health condition, and each item is answered yes or no.

CONTACTS AND LOCATIONS:
Locations (1):
- Ufuk University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided